CLINICAL TRIAL: NCT05364606
Title: Patient Specific Talus Spacer Post Approval Study
Status: Recruiting | Type: Observational
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: AOPSTSPAS
Record Dates: First submitted 2022-02-04; First posted 2022-05-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Avascular Necrosis of the Talus
Keywords: Avascular Necrosis; Talus; Ankle
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 50 Subjects: 50 Subjects Receiving the Patient Specific Talus Spacer.
  Interventions: Device: Patient Specific Talus Spacer

INTERVENTIONS:
Device: Patient Specific Talus Spacer — Patient Specific Talus Spacer is a solid polished replica of the patient's bone.

SUMMARY:
Humanitarian Device Exemption Approved Patient Specific Talus Spacer Post Approval Study.

DETAILED DESCRIPTION:
This is a Humanitarian Device Exemption (HDE) approved device called the Patient Specific Talus Spacer. This is a post approval study to determine the safety and probable benefit of the Patient Specific Talus Spacer in commercial use. The Patient Specific Talus Spacer is a solid polished replica of the patient's bone to allow the patient to regain motion and reduce pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject plans to undergo implantation of the Patient Specific Talus Spacer for avascular necrosis of the ankle joint independent of this research protocol;
2. Avascular necrosis of the ankle joint;
3. Age 21 years old or older;
4. Subject has good general health; and
5. Subject signs a written informed consent form (ICF) prior to the surgical procedure.

Exclusion Criteria:

1. Presence of any contraindication identified in the device Instructions for Use;
2. Surgeon determines that the patient is not appropriate for the Talus Spacer procedure based on the device IFU (including the enumerated Warnings and Precautions);
3. Based on the medical opinion of the surgeon, the patient is not appropriate for the Talus Spacer procedure;
4. For female subjects, pregnancy;
5. Active systemic disease, such as AIDS, HIV, or active infection;
6. Active infection or the skin is compromised at the surgical site; and
7. Systemic disease that would affect the subject's welfare;
8. Is a prisoner, incarcerated, or has been coerced to participate in the study that could impact the validity of results;
9. Is currently participating in an investigational therapy (device and/or pharmaceutical) within 30 days prior to entering the study or such treatment is planned during the time course of follow-up.
10. If the Sponsor has notified the site that 30 subjects have been enrolled in the study with a Cobalt Chromium Patient Specific Talus Spacer, and the surgeon believes that a Cobalt Chromium Patient Specific Talus Spacer is the best option for the patient.
11. If the Sponsor has notified the site that 30 subjects have been enrolled in the study with a Titanium (Ti6Al4V) with Titanium Nitride (TiN) coating Patient Specific Talus Spacer, and the surgeon believes that a Titanium (Ti6Al4V) with Titanium Nitride (TiN) coating Patient Specific Talus Spacer is the best option for the patient.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Avascular Necrosis of the Ankle Joint.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinically Significant Improvement in Pain on the Visual Analog Scale (VAS) | At 5 years compared to Baseline
  Clinically Significant Improvement in Pain on the Visual Analog Scale (VAS) at 5 years compared to baseline on the 0 to 100mm scale. A lower score will indicate an improvement in pain.
A lack Secondary Subsequent Surgical Intervention at 5 years Post Operative assessed during the subject's visits | A patient will achieve the primary probable benefit endpoint only is they do not undergo a Secondary Subsequent Surgical Intervention at 5 years Post Operative as assessed during the subjects visits for the study.
  A lack Secondary Subsequent Surgical Intervention (SSSI) at 5 years Post Operative

SECONDARY OUTCOMES:
Additional Analyses at 5 years Post Operative compared to baseline, Range of Motion of the Ankle. | 5 Years Post Procedure compared to baseline.
  Additional analyses will be performed to observe improvement at 5-years post-procedure compared to baseline on ankle range of motion (ROM) as assessed by the surgeon at each follow up visit through 5 years Post Operative.

OTHER OUTCOMES:
Additional Analyses at 5 Years Post Operative compared to Baseline for Foot and Outcome Score FAOS | 5 Years Post Procedure compared to baseline
  Additional analyses will be performed to observe improvement at 5-years post-procedure compared to baseline on Foot and Ankle Outcome Score (FAOS - which include Pain, Other Symptoms, Sport and Recreation Function, Activities of Daily Living (ADL) and Foot and Ankle related Quality of Life (QOL). This is a series of questions for each sub section that the subject will answer at the subjects visits.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Redwood Orthopaedics, Santa Rosa, California
  - Fort Wayne Orthopedics, Fort Wayne, Indiana
  - Mercy Institute for Foot & Ankle Reconstruction, Baltimore, Maryland
  - Duke Orthopeadics Arringdon, Morrisville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Physicians Orthopedics - Pearland, Pearland, Texas

IPD SHARING:
Plan to Share IPD: Undecided
After study completion and data analysis, results of the study will be shared with the Investigator's who participated. Individual Patient Identifiers will not be provided. Only specific numbers from the statistical analysis will be shared.